CLINICAL TRIAL: NCT03053362
Title: An Open-Label Clinical Trial Evaluating Sensitivity to Change in Cognition Using the THINC-it Following Treatment With Vortioxetine in Major Depressive Disorder
Brief Title: THINC-it Vortioxetine - Sensitivity to Change
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Brain and Cognition Discovery Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00020418
Record Dates: First submitted 2017-02-07; First posted 2017-02-15 (Actual); Results first posted 2022-01-20 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Major Depressive Disorder; Cognitive Change
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine

STUDY DESIGN:
Intervention Model Description: Determining the effectiveness of a new tool used to detect changes in cognition among individuals with MDD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Major Depressive Disorder Population (Experimental): 100 Individuals with DSM-5-defined MDD, aged 18-65
  All participants receiving vortioxetine for a total of 8 weeks. Participants will receive10 mg/day on days 1-14 of the study treatment period, with the option to increase to vortioxetine 20 mg/day at the end of Week 2 based on physician's judgment. For the remaining 6 weeks, the dose of vortioxetine will be flexible at 10 or 20 mg/day as decided by a research doctor.
  Patients will receive the THINC-it over 3 time frame periods. The THINC-it comprised of: Spotter, Symbol Check, Codebreaker, Trails, and PDQ-5-D.
  Interventions: Drug: Vortioxetine; Other: THINC-it Tool
- Healthy Control Population (Other): 50 Healthy Controls (18-65 years of age) matched on sex, age, and years of education
  Interventions: Other: THINC-it Tool

INTERVENTIONS:
Drug: Vortioxetine — Observing change in cognition using THINC-it tool in patients with MDD.
  Arms: Major Depressive Disorder Population
Other: THINC-it Tool — Digitalized cognitive test application administering the following cognitive test components:
  Digit Symbol Substitution Test (DSST) Choice Reaction Time (CRT) One-back working memory tool Trail Making Test B (TMT-B) Perceived Deficits Questionnaire-5 Depression (PDQ-5-D)

SUMMARY:
The purpose of this study is to evaluate the sensitivity of the THINC-it tool, in measuring change in cognitive deficits in individuals with MDD after receiving vortioxetine.

DETAILED DESCRIPTION:
Vortioxetine is used in this study as an antidepressant to improve mood, cognition and quality of life. "Cognition" refers to intellectual functions such as thinking, understanding, learning and remembering. Vortioxetine is approved by Health Canada for the treatment of MDD. In addition, vortioxetine has been reported to have a beneficial effect on cognitive areas such as executive function, attention/speed of processing, and memory, that are commonly affected negatively by MDD. Vortioxetine is recognized by Health Authorities in the EU and many other countries as having a benefit on cognitive dysfunction (loss of intellectual functions) in patients with MDD.Cognitive dysfunction is a highly persistent, pervasive and progressive abnormality in young adults (i.e., 18-65 years) with MDD.

It has also been shown that among adults with MDD who are gainfully employed, measures of cognition are a greater determinant of overall workplace performance than is total depression symptom severity. Several lines of evidence indicate that cognitive deficits that persist between episodes of depression are critical determinants of functional recovery in the workplace. The functional implications associated with cognitive impairment provide the impetus for systematic evaluation, measurement and assessment of the domains of cognition expected to be impaired in this patient population.

To date, no measurement tool has been sufficiently validated and/or determined to be sensitive to the cognitive deficits in younger adults with MDD. Major limitations of available comprehensive psychometric tools include relative lack of availability, cost, lack of access to most healthcare providers, and above all else, the lengthy time to administer. Moreover, the need for a psychometrist to interpret the results adds to the complexity and the costliness of such an endeavor.

It is imperative that any tool recommended for clinical utility be aligned with the busy nature of a high-volume clinical practice. The ideal gold standard tool for assessing the presence of cognitive dysfunction in MDD in the clinical environment should include, but not be limited to, features such as good conceptual coverage of cognitive domains affected in MDD, good sensitivity and reliability, and it should be relatively uninfluenced by culture effects and practice effects. The tool would also need to be brief, easy to administer and interpret, and complement busy clinical practice.

It is anticipated that the THINC-it tool will be free of charge and downloadable from the THINC-it website for use in the primary care and specialty setting. The THINC-it tool will be accessible via computers/tablets, will take 20 minutes to self-administer in a clinical setting, and the performance results will be immediately available.

ELIGIBILITY:
MDD Population

Inclusion Criteria:

1. The participant is able and willing to provide informed consent.
2. The participant is male or female 18-65 years of age.
3. The participant has received a current diagnosis of a major depressive episode (MDE) as part of MDD as per DSM-5 criteria.
4. The participant's current MDE is confirmed by the Mini International Neuropsychiatric Interview (M.I.N.I 5.0.).
5. The participant is an outpatient of a psychiatric setting.
6. The participant has a MADRS score ≥ 26 at screening and baseline.
7. The participant's reported duration of the current MDE is at least 3 months.
8. At least one prior major depressive episode validated by previous treatment (e.g., guideline-informed pharmacotherapy and/or manual-based psychotherapy).
9. All participants will be screened for cognitive impairment based on DSST performance (pen-and-paper version) with a maximum baseline score of 70 correct symbols entered to avoid ceiling effects.

Exclusion Criteria:

1. Current alcohol and/or substance use disorder.
2. Presence of comorbid psychiatric disorder other than MDD that is a focus of clinical concern as confirmed by the M.I.N.I 5.0.
3. Medications approved and/or employed off-label for cognitive dysfunction (e.g., psychostimulants).
4. Any medication for a general medical disorder that, in the opinion of the investigator, may affect cognitive function (e.g., corticosteroids, beta-blockers).
5. Use of benzodiazepines within 12 hours of cognitive assessments.
6. Consumption of alcohol within 8 hours of cognitive assessments.
7. Recent use of marijuana as determined by a toxicology screen.
8. Physical, cognitive, or language impairments sufficient to adversely affect data derived from cognitive assessments.
9. Diagnosis reading disability or dyslexia.
10. Clinically significant learning disorder by history.
11. Electroconvulsive therapy (ECT) in the last 6 months.
12. History of moderate or severe head trauma (e.g., loss of consciousness for >1 hour), other neurological disorders, or unstable systemic medical diseases that in the opinion of the investigator are likely to affect the central nervous system.
13. Pregnant and/or breastfeeding.
14. Received investigational agents as part of a separate study within 30 days of the screening visit.
15. Actively suicidal or evaluated as being a suicide risk (a score of > 4 on the MADRS and/or per clinical judgment using the Columbia-Suicide Severity Rating Scale).
16. Currently receiving treatment with Monoamine Oxidase Inhibitors (MAOIs) anti-depressants, antibiotics such as linezolid, or intravenous methylene blue.

Healthy Control Population

Inclusion Criteria:

1. No current or past history of mental disorder as evidenced by the M.I.N.I. 5.0 for DSM-IV.
2. No first-degree relative with an established diagnosis by a healthcare provider of a mood or psychiatric disorder.
3. No unstable medical disorders.

Exclusion Criteria:

1. Use of any medication for a general medical disorder and/or condition that, in the opinion of the investigator, may affect cognitive function (e.g., corticosteroids, beta-blockers).
2. Pregnant and/or breastfeeding.
3. Consumption of alcohol within 8 hours of THINC-it tool administration.
4. Recent use of marijuana as determined by a toxicology screen.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2018-08-08 (Actual); Study Completion 2018-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger McIntyre, Principal Investigator — Brain and Cognition Discovery Foundation
Locations (1):
- CRTCE/KJK Healthplex, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McIntyre RS, Subramaniapillai M, Park C, Zuckerman H, Cao B, Lee Y, Iacobucci M, Nasri F, Fus D, Bowie CR, Tran T, Rosenblat JD, Mansur RB. The THINC-it Tool for Cognitive Assessment and Measurement in Major Depressive Disorder: Sensitivity to Change. Front Psychiatry. 2020 Jun 24;11:546. doi: 10.3389/fpsyt.2020.00546. eCollection 2020. PMID 32670103
- [Derived] Subramaniapillai M, Mansur RB, Zuckerman H, Park C, Lee Y, Iacobucci M, Cao B, Ho R, Lin K, Phan L, McIntyre RS. Association between cognitive function and performance on effort based decision making in patients with major depressive disorder treated with Vortioxetine. Compr Psychiatry. 2019 Oct;94:152113. doi: 10.1016/j.comppsych.2019.07.006. Epub 2019 Jul 24. PMID 31404802
- [Derived] Cao B, Park C, Subramaniapillai M, Lee Y, Iacobucci M, Mansur RB, Zuckerman H, Phan L, McIntyre RS. The Efficacy of Vortioxetine on Anhedonia in Patients With Major Depressive Disorder. Front Psychiatry. 2019 Jan 31;10:17. doi: 10.3389/fpsyt.2019.00017. eCollection 2019. PMID 30766492

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Healthy volunteers were recruited on an ongoing basis until 50 completed volunteers were enrolled. Eight participants began the study but did not complete the study.
Groups:
- Major Depressive Disorder Population: 100 Individuals with DSM-5-defined MDD, aged 18-65
  All participants receiving vortioxetine for a total of 8 weeks. Participants will receive10 mg/day on days 1-14 of the study treatment period, with the option to increase to vortioxetine 20 mg/day at the end of Week 2 based on physician's judgment. For the remaining 6 weeks, the dose of vortioxetine will be flexible at 10 or 20 mg/day as decided by a research doctor.
  Patients will receive the THINC-it over 3 time frame periods. The THINC-it comprised of: Spotter, Symbol Check, Codebreaker, Trails, and PDQ-5-D.
  Vortioxetine: Observing change in cognition using THINC-it tool in patients with MDD.
  THINC-it Tool: Digitalized cognitive test application administering the following cognitive test components:
  Digit Symbol Substitution Test (DSST) Choice Reaction Time (CRT) One-back working memory tool Trail Making Test B (TMT-B) Perceived Deficits Questionnaire-5 Depression (PDQ-5-D)
- Healthy Control Population: 50 Healthy Controls (18-65 years of age) matched on sex, age, and years of education
  THINC-it Tool: Digitalized cognitive test application administering the following cognitive test components:
  Digit Symbol Substitution Test (DSST) Choice Reaction Time (CRT) One-back working memory tool Trail Making Test B (TMT-B) Perceived Deficits Questionnaire-5 Depression (PDQ-5-D)
Period: Overall Study
Arm/Group | Major Depressive Disorder Population | Healthy Control Population
Started | 100 | 58
Completed | 83 | 50
Not Completed | 17 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Major Depressive Disorder Population | Healthy Control Population | Total
Number analyzed (Participants) | 100 | 58 | 158
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.90 (12.74) | 43.00 (13.89) | 40.41 (13.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 27 | 94
  Male | 33 | 31 | 64
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 68 | 20 | 88
  Asian | 11 | 16 | 27
  Other | 21 | 22 | 43
Region of Enrollment [Number; unit: participants]
  Canada | 100 | 58 | 158
Baseline Montgomery Åsberg Depression Rating Scale (MADRS) [Mean (Standard Deviation); unit: units on a scale] — Changes in mood assessed by the Montgomery Åsberg Depression Rating Scale [MADRS]. The overall score ranges from 0 to 60, where greater scores indicate worse depression.
  units on a scale | 31.83 (7.54) | 1.64 (2.41) | 20.75 (5.66)
Baseline Digit Symbol Substitution Task Total Score (DSST) [Mean (Standard Deviation); unit: units on a scale] — The measure assesses the number of correct symbols copied by the participants. Higher scores indicate better performance (lowest score 0 and highest score is 133)
  units on a scale | 56.05 (14.70) | 61.21 (14.25) | 57.94 (14.53)
Baseline Trail Making Test - Part B (TMT-B) [Mean (Standard Deviation); unit: time (seconds)] — Cognition assessed by the TMT-B. The outcome measure is time in seconds, where greater time indicates worse performance.
  time (seconds) | 72.94 (30.59) | 70.59 (29.14) | 72.08 (30.06)
Baseline THINC-it Tool Objective z-score [Mean (Standard Deviation); unit: z-score] — Change in cognition as measured by the objective assessments of cognition within the THINC-it tool. "THINC-it" is the name of the cognition tool and is not an acronym. The objective measurements that comprise the THINC-it tool include the Spotter task (Choice Reaction Time), Symbol Check task(1-back test),Trails task(Trails Making Test B), and Codebreaker task (Digit Symbol Substitution Test). The composite score from all four tests were converted to standard z-score. Higher z-scores indicate better cognition. A z-score of zero represents the population mean.
  z-score | -0.05 (0.76) | -0.12 (0.82) | -0.08 (0.78)

OUTCOME MEASURES:

1. Primary Outcome: Cognition Measured Using the THINC-it Tool
Description: Change in cognition as measured by the objective assessments of cognition within the THINC-it tool. "THINC-it" is the name of the cognition tool and is not an acronym. The objective measurements that comprise the THINC-it tool include the Spotter task (Choice Reaction Time), Symbol Check task(1-back test),Trails task(Trails Making Test B), and Codebreaker task (Digit Symbol Substitution Test). The composite score from all four tests were converted to standard z-score. Higher z-scores indicate better cognition. A z-score of zero indicates population mean.
Time Frame: Baseline and 8 weeks
Population: Participants were either lost to follow up or dropped out of the study.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Major Depressive Disorder Population | Healthy Control Population
Number analyzed (Participants) | 100 | 58
z-score
  Week 0 | -0.05 (0.76) | -0.12 (0.82)
  Week 8: number analyzed (Participants) | 83 | 50
  Week 8 | 0.12 (0.73) | 0 (0.77)

2. Secondary Outcome: Changes in Mood as Measured by the Montgomery Åsberg Depression Rating Scale (MADRS)
Description: Changes in mood assessed by the Montgomery Åsberg Depression Rating Scale [MADRS]. The overall score ranges from 0 to 60, where greater scores indicate worse depression.
Time Frame: Baseline and 8 weeks
Population: Participants dropped out or lost to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Healthy Control Participants: 50 age, and sex-matched healthy controls who did not meet DSM-5 criteria for major depressive disorder
Arm/Group | Major Depressive Disorder Population | Healthy Control Participants
Number analyzed (Participants) | 99 | 58
units on a scale
  Week 0 | 31.83 (7.54) | 1.64 (2.41)
  Week 8: number analyzed (Participants) | 82 | 47
  Week 8 | 20.39 (10.66) | 1.02 (1.78)

3. Secondary Outcome: Changes in Cognitive Function Assessed by the Digit Symbol Substitution Task (DSST)
Description: Changes in cognition assessed by the Digit Symbol Substitution Task (DSST). The outcome measure is the number of correct symbols copied by the participants. Higher scores indicate better performance (minimum score is 0 and maximum is 133).
Time Frame: Baseline and 8 weeks
Population: Participants dropped out or lost to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Major Depressive Disorder Population | Healthy Control Participants
Number analyzed (Participants) | 100 | 58
units on a scale
  Week 0 | 56.05 (14.70) | 61.21 (14.27)
  Week 8 | 64.14 (14.84) | 67.53 (14.14)

4. Secondary Outcome: Changes in Cognitive Function Assessed by the Trail Making Test - Part B (TMT-B)
Description: Changes in cognition assessed by the TMT-B. The outcome measure is time in seconds, where greater time indicates worse performance.
Time Frame: Baseline and 8 weeks
Population: Participants dropped out or lost to follow-up.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Major Depressive Disorder Population | Healthy Control Participants
Number analyzed (Participants) | 99 | 58
seconds
  Week 0 | 72.95 (30.60) | 70.60 (29.14)
  Week 8: number analyzed (Participants) | 83 | 49
  Week 8 | 62.72 (40.50) | 58.71 (21.08)

5. Secondary Outcome: Changes in Global Functional Impairment Using the Sheehan Disability Scale Total Score
Description: Sheehan Disability Scale rates the extent to which his or her 1) work, 2) social life or leisure activities, and 3) home life or family responsibilities are impaired by his or her symptoms on a 10-point visual analog scale. The numerical ratings of 0-10 can be translated into a percentage if desired. The three items may be summed into a single dimensional measure of global functional impairment that ranges from 0 (unimpaired) to 30 (highly impaired).
Time Frame: Baseline and 8 weeks
Population: Participants dropped out or lost to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Major Depressive Disorder Population | Healthy Control Participants
Number analyzed (Participants) | 100 | 56
units on a scale
  Week 0 | 20.63 (6.10) | 0.98 (2.93)
  Week 8 | 14.64 (8.48) | 1.3 (4.35)

6. Secondary Outcome: Changes in the World Health Organization Wellbeing Index (5-Item)
Description: The WHO-5 is a short questionnaire consisting of 5 simple and non-invasive questions, which tap into the subjective well-being of the respondents. The WHO-5 only contains positively phrased items. The respondent is asked to rate how well each of the 5 statements applies to him or her when considering the last 14 days. Each of the 5 items is scored from 5 (all of the time) to 0 (none of the time). The raw score therefore theoretically ranges from 0 (absence of well-being) to 25 (maximal well-being). A percent score out of 25 is reported.
Time Frame: Baseline and 8 weeks
Population: Participants dropped out or lost to follow-up.
Measure: Mean (Standard Deviation); unit: percent of maximum score
Arm/Group | Major Depressive Disorder Population | Healthy Control Participants
Number analyzed (Participants) | 100 | 57
percent of maximum score
  Week 0 | 15.24 (11.45) | 72.42 (16.42)
  Week 8: number analyzed (Participants) | 83 | 57
  Week 8 | 29.16 (20.35) | 73.60 (17.22)

7. Secondary Outcome: Changes in Changes in Anhedonia From Baseline to Week 8
Description: To establish sensitivity to change in anhedonia using the Snaith-Hamilton Pleasure Scale (SHAPS) total score in adults (18-65) with MDD treated with vortioxetine (10-20 mg flexibly dosed for 8 weeks). The SHAPS total score in adults ranges from 14 to 56. Higher score indicates more pleasure, with maximum of 56 points on the scale.
Time Frame: Baseline and 8 weeks
Population: Participants dropped out or lost to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Major Depressive Disorder Population | Healthy Control Participants
Number analyzed (Participants) | 99 | 57
units on a scale
  Week 0 | 35.12 (6.74) | 51.12 (4.53)
  Week 8: number analyzed (Participants) | 83 | 50
  Week 8 | 40.33 (7.49) | 50.38 (4.76)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the 8-week trial from baseline to endpoint.
Description: At each visit, participants were asked if they experienced any health problems or side effects since the previous visit. All adverse events (AE) were recorded appropriately, whether or not considered related to vortioxetine. This included AEs spontaneously reported by the participant and/or observed by members of the research team as well as AEs reported in response to a direct question (e.g. "Have you experienced any health problems or side effects since your last visit?")
Arm/Group | Major Depressive Disorder Population | Healthy Control Population
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/50
Other Adverse Events (participants affected / at risk) | 53/100 | 0/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Major Depressive Disorder Population (N=100) | Healthy Control Population (N=50)
Nausea (Gastrointestinal disorders) | 42 (42) | 0 (0) — Variable degree and duration of nausea experienced by participants with major depression taking vortioxetine. This was an expected side effect of the medication.
Vomiting (Gastrointestinal disorders) | 5 (5) | 0 (0)
Gastrointestinal Upset (Gastrointestinal disorders) | 16 (16) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (6) | 0 (0)
Headache (Nervous system disorders) | 15 (15) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 0 (0)
Dizziness/Lightheadedness (Nervous system disorders) | 13 (13) | 0 (0)
Itchiness (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-08): https://cdn.clinicaltrials.gov/large-docs/62/NCT03053362/Prot_SAP_000.pdf
  • Informed Consent Form (2017-11-10): https://cdn.clinicaltrials.gov/large-docs/62/NCT03053362/ICF_001.pdf